CLINICAL TRIAL: NCT02029521
Title: Supplementation of Oral Reduced Glutathione in Pediatric Cystic Fibrosis for Growth Failure
Brief Title: Supplementation of Oral Reduced Glutathione in Pediatric Cystic Fibrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clark Bishop (Other)
Responsible Party: Sponsor-Investigator, Clark Bishop, Co investigator, Brigham Young University
Organization: Brigham Young University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIMP/clin.stud/2010/1.
Record Dates: First submitted 2013-12-30; First posted 2014-01-08 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; growth Failure; glutathione
MeSH Terms: conditions — Cystic Fibrosis; Failure to Thrive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral reduced l-glutathione (Experimental): The treatment was pharmaceutical-grade Reduced L-Glutathione (GSH) with a daily dose of 65 mg/kg.
  Interventions: Dietary Supplement: Oral reduced l-glutathione
- Placebo Calcium Citrate (Placebo Comparator): The placebo was calcium citrate with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Oral reduced l-glutathione — The treatment was pharmaceutical-grade Reduced L-Glutathione (GSH) with a daily dose of 65 mg/kg. The placebo was calcium citrate with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
  Arms: Oral reduced l-glutathione
Dietary Supplement: Placebo — calcium citrate with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
  Arms: Placebo Calcium Citrate

SUMMARY:
Many individuals with cystic fibrosis experience growth failure. The reasons are not clear, but inflammation of the gut in these patients seems to be one important reason. Glutathione is important to normal function of the intestine and lungs. Glutathione functions to decrease inflammation and to thin mucus. However, in cystic fibrosis, glutathione gets trapped inside of cells, so it cannot travel to the surface of the cells and perform its proper function. Moreover, glutathione has been shown to improve nutritional status in patients with AIDS and cancer.

Investigators hypothesize that supplementation of oral glutathione to pediatric individuals with cystic fibrosis could improve growth failure.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is known principally for its pulmonary consequences. However, for most individuals with CF, the earliest manifestations are not pulmonary, but gastro-intestinal. Many children experience growth failure. Chronic gut inflammation also develops. Research has also established that lung function scores are significantly correlated with Body Mass Index (BMI) and weight percentile in CF. Therefore, interventions to improve the gastro-intestinal dimension of CF in early childhood have the potential to ameliorate the course of the disease over the life span of the patient. Both Cochrane Database reviews and a recent review commissioned by the Cystic Fibrosis Foundation found only fair evidence for current nutritional guidelines.Therefore, there is a pressing need for a treatment for CF growth failure that is more effective and less invasive than current treatments.

The discovery that CF is associated with significantly diminished efflux of reduced glutathione (GSH) from most cells in the body offers a new perspective on the pathophysiology of this disease. GSH plays several important roles; among the most important are the following: 1) primary water-soluble antioxidant; 2) mucolytic capable of cleaving disulfide bonds; and 3) regulator of immune system function. The relationship between redox ratio (GSH:GSSG) and total glutathione (GSH+GSSG) and the initiation of inflammation is well established in the research literature.

GSH is also an important component of the epithelial lining fluid of the intestines, helping to keep intestinal mucus thin, serving to defend the intestinal system against reactive oxygen species, and keeping inflammation in check under normal circumstances. GSH is an FDA-approved treatment for AIDS-related cachexia. The growing recognition of GSH system dysfunction in CF, coupled with an established research literature on the role of GSH in gastro-intestinal function and weight gain in non-CF contexts, suggest a new intervention for growth failure in early childhood in CF patients. Specifically, investigators hypothesized that oral glutathione could effectively treat CF growth failure in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of Cystic Fibrosis by either of the following criteria: >60 sweat chloride test or paired deleterious DNA cystic fibrosis transmembrane conductance regulator (CFTR) mutations (Ambry genetics, Genetech or ARUP);

-Pancreatic insufficient as defined by doctor's prescription of pancreatic enzymes.

Exclusion Criteria:

* Hospitalized for bowel obstruction or surgery in the six months prior to enrollment;
* had had a pulmonary exacerbation or oral steroid use or IV antibiotics within one month of enrollment,
* who had been taking either GSH or N-acetyl cysteine (NAC) within the 12 month period immediately prior to the trial,
* chronically infected with Burkholderia cepacia.

Ages: 18 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clark T Bishop, MD, Study Director — Intermountain Health Care
Locations (1):
- Turin, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Reduced L-glutathione: The treatment was pharmaceutical-grade Reduced L-Glutathione (GSH) with a daily dose of 65 mg/kg.
  Oral reduced l-glutathione: The treatment was pharmaceutical-grade Reduced L-Glutathione (GSH) with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
Period: Overall Study
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Started | 24 | 23
Completed | 22 | 22
Not Completed | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Pediatric cystic fibrosis patients, ages 15 months to 10 years
Groups:
- Oral Reduced L-glutathione: The treatment was pharmaceutical-grade Reduced L-Glutathione (GSH) with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
- Placebo Oral Calcium Citrate: The placebo was calcium citrate with a daily dose of 65 mg/kg. The daily dose of each substance was divided into three doses given at mealtime.
- Total: Total of all reporting groups
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Customized [Number; unit: participants] — 15 months to 3 years and greater than 3 years
  participants
    15 months to 3 years | 6 | 6 | 12
    3 years to 10 years | 16 | 16 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 8 | 12 | 20
Region of Enrollment [Number; unit: participants]
  Italy | 22 | 22 | 44
Body Mass Index Percentile [Mean (Standard Deviation); unit: Percentile adjusted for age and sex] — Body Mass Index for patients with standardized percentile
  Percentile adjusted for age and sex | 25.1 (15.9) | 31.1 (14.1) | 28.3 (15.1)
Weight Percentile [Mean (Standard Deviation); unit: Percentile adjusted for sex and age] | 24.2 (13.7) | 33.5 (13.4) | 26.9 (13.6)
Height Percentile [Mean (Standard Deviation); unit: Percentile adjusted for weight and heigh] | 36.3 (14.4) | 39.3 (13.5) | 37.7 (13.9)
Fecal Calprotectin [Mean (Standard Deviation); unit: micrograms/gram feces] | 113.2 (52.5) | 76.1 (32.2) | 94.6 (47)
Forced Expiratory Volume at one second. [Mean (Standard Deviation); unit: Percent predicted] — Forced Expiratory Volume at one second. Percentile normalized by age, height and gender.
  Percent predicted | 63.5 (4.8) | 71 (7.8) | 66.9 (7.3)
Forced Vital Capacity [Mean (Standard Deviation); unit: Percent Predicted] — Forced Vital Capacity percentile normalized by age, height and gender
  Percent Predicted | 81.8 (8.7) | 88.2 (9.6) | 84.7 (9.4)
Gene Mutations [Number; unit: participants]
  G551D/1303K | 1 | 0 | 1
  DelF508/R117H | 1 | 0 | 1
  R117H/G542X | 1 | 2 | 3
  DelF508/DelF508 | 4 | 5 | 9
  DelF508/R553X | 2 | 0 | 2
  W1282X/R347P | 1 | 0 | 1
  DelF508/N1303K | 1 | 1 | 2
  DelF508/3849+10KBCT | 1 | 1 | 2
  G551D/621+1GT | 1 | 0 | 1
  W1282X/DelF508 | 2 | 1 | 3
  R117H/R347P | 1 | 1 | 2
  R117H/W1282X | 1 | 0 | 1
  DelF508/G542X | 1 | 2 | 3
  3849+10kb/N1303k | 1 | 0 | 1
  N1303K/R553X | 1 | 0 | 1
  G551D/DelF508 | 1 | 2 | 3
  R117H/1466delAATT | 1 | 0 | 1
  DelF508/G576X | 0 | 1 | 1
  DelF508/S489X | 0 | 1 | 1
  G542X/G542X | 0 | 1 | 1
  DelF508/R347P | 0 | 1 | 1
  R117H/R117H | 0 | 1 | 1
  N1303k/G542X | 0 | 2 | 2
Sweat Chloride Test [Mean (Standard Deviation); unit: mmol/L] | 87.7 (15.8) | 85.0 (15.6) | 86.3 (15.6)
Participants' Lipase Intake in Units Per Day [Mean (Standard Deviation); unit: units of lipase] | 130909.1 (54590.2) | 123181.8 (47044.7) | 127045.5 (50512.7)
Bacteriology [Number; unit: participants]
  A. xylososidans | 3 | 1 | 4
  MRSA | 0 | 1 | 1
  PA | 2 | 3 | 5
  Staph | 7 | 9 | 16
  Normal flora | 3 | 2 | 5
  PA and S. maltophilia | 1 | 0 | 1
  PA and Staph | 5 | 6 | 11
  Staph and A. xylososidans | 1 | 0 | 1
White Blood Cell Count [Mean (Standard Deviation); unit: 1000 cells/mm^3] — Total White Blood Cell Count. 1000 per cubic millimeter
  1000 cells/mm^3 | 9.1 (2.0) | 8.9 (2.7) | 9.0 (2.4)
ALT [Mean (Standard Deviation); unit: units per liter] — peripheral blood Alanine AminoTransferase
  units per liter | 23.2 (9.3) | 22.6 (11.4) | 22.9 (10.3)
Vitamin E [Mean (Standard Deviation); unit: micrograms per ml.] — Peripheral blood vitamin E, micrograms per ml.
  micrograms per ml. | 7.7 (1.6) | 7.5 (1.6) | 7.6 (1.6)
C-Reactive Protein [Mean (Standard Deviation); unit: miligrams per liter] — C-Reactive Protein in peripheral blood
  miligrams per liter | 13.3 (7.7) | 12.1 (6.6) | 12.7 (7.1)
Frequency of Abdominal Pain [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 7 | 11 | 18
    2- rare | 10 | 4 | 14
    3- frequently | 4 | 6 | 10
    4- constantly | 1 | 1 | 2
Severity of Abdominal Pain [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 6 | 11 | 17
    2- light | 12 | 4 | 16
    3- moderate | 3 | 7 | 10
    4- serious | 1 | 0 | 1
Frequency of Belching [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 14 | 15 | 29
    2- rare | 3 | 3 | 6
    3- frequently | 5 | 4 | 9
    4- constantly | 0 | 0 | 0
Severity of Belching [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 14 | 3 | 17
    2- light | 5 | 10 | 15
    3- moderate | 3 | 8 | 11
    4- serious | 0 | 1 | 1
Frequency of Flatulence [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 3 | 4 | 7
    2- rare | 10 | 9 | 19
    3- frequently | 8 | 9 | 17
    4- constantly | 1 | 0 | 1
Severity of Flatulence [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 3 | 4 | 7
    2- light | 11 | 10 | 21
    3- moderate | 8 | 8 | 16
    4- serious | 0 | 0 | 0
Frequency of Lack of Appetite [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 1 | 5 | 6
    2- rare | 10 | 13 | 23
    3- frequently | 8 | 4 | 12
    4- constantly | 3 | 0 | 3
Severity of Lack of Appetite [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 1 | 5 | 6
    2- light | 11 | 13 | 24
    3- moderate | 7 | 4 | 11
    4- serious | 3 | 0 | 3
Frequency of Bloating [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 2 | 4 | 6
    2- rare | 7 | 7 | 14
    3- frequently | 12 | 10 | 22
    4- constantly | 1 | 1 | 2
Severity of Bloating [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 2 | 4 | 6
    2- light | 7 | 7 | 14
    3- moderate | 13 | 10 | 23
    4- serious | 0 | 1 | 1
Frequency of Nausea [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 11 | 15 | 26
    2- rare | 8 | 7 | 15
    3- frequently | 3 | 0 | 3
    4- constantly | 0 | 0 | 0
Severity of Nausea [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 11 | 15 | 26
    2- light | 9 | 6 | 15
    3- moderate | 2 | 1 | 3
    4- serious | 0 | 0 | 0
Frequency of Vomiting [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 16 | 18 | 34
    2- rare | 6 | 4 | 10
    3- frequently | 0 | 0 | 0
    4- constantly | 0 | 0 | 0
Severity of Vomiting [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 16 | 18 | 34
    2- light | 6 | 4 | 10
    3- moderate | 0 | 0 | 0
    4- serious | 0 | 0 | 0
Frequency of Heart Burn [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 17 | 18 | 35
    2- rare | 1 | 2 | 3
    3- frequently | 4 | 2 | 6
    4- constantly | 0 | 0 | 0
Severity of Heart Burn [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 17 | 18 | 35
    2- light | 1 | 1 | 2
    3- moderate | 4 | 3 | 7
    4- serious | 0 | 0 | 0
Frequency of Diarrhea [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 9 | 9 | 18
    2- rare | 9 | 11 | 20
    3- frequently | 4 | 2 | 6
    4- constantly | 0 | 0 | 0
Severity of Diarrhea [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 9 | 10 | 19
    2- light | 10 | 10 | 20
    3- moderate | 3 | 2 | 5
    4- serious | 0 | 0 | 0
Frequency of More than 2 Bowel Movements Per Day [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 4 | 10 | 14
    2- rare | 12 | 6 | 18
    3- frequently | 5 | 6 | 11
    4- constantly | 1 | 0 | 1
Severity of More Than 2 Bowel Movements Per Day [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 4 | 10 | 14
    2- light | 12 | 8 | 20
    3- moderate | 5 | 4 | 9
    4- serious | 1 | 0 | 1
Frequency of Less Than 2 Bowel Movements Per Week [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
  participants
    1- never | 18 | 17 | 35
    2- rare | 0 | 2 | 2
    3- frequently | 4 | 3 | 7
    4- constantly | 0 | 0 | 0
Severity of Less Than 2 Bowel Movements Per Week [Number; unit: participants] — Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
  participants
    1- absent | 18 | 17 | 35
    2- light | 0 | 3 | 3
    3- moderate | 4 | 2 | 6
    4- serious | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Weight Percentile at 3 Months
Description: Weight Percentile at 3 months adjusted for sex and age
Time Frame: 3 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: Weight Percentile, sex and age adjusted
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
Weight Percentile, sex and age adjusted | 33.5 (14.9) | 31.0 (13.4)

2. Primary Outcome: Height Percentile
Description: Height Percentile adjusted for sex and age
Time Frame: 3 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: Percentile adjusted for age and sex
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
Percentile adjusted for age and sex | 39.3 (11.9) | 38.0 (13.8)

3. Primary Outcome: BMI Percentile
Description: Body Mass Index percentile adjusted for sex and age. Standard BMI are not available for participants under 2 years of age
Time Frame: 3 months
Population: BMI percentile not available for children under 2 years of age.
Measure: Mean (Standard Deviation); unit: Percentile adjusted for age and sex
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 20 | 20
Percentile adjusted for age and sex | 37.1 (33.6) | 47.5 (17.0)

4. Secondary Outcome: Forced Vital Capacity
Description: Forced vital capacity percent predicted
Time Frame: 3 months
Population: Pulmonary function tests not performed on children under the age of 5
Measure: Mean (Standard Deviation); unit: percent predicted
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 11 | 9
percent predicted | 87.2 (7.2) | 88.8 (10.3)

5. Secondary Outcome: FEV1
Description: Forced expiratory volume at one second, percent predicted
Time Frame: 3 months
Population: Pulmonary function tests not performed on children under the age of 5
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 11 | 9
Percent predicted | 73.2 (5.6) | 73.0 (11.1)

6. Secondary Outcome: Bacteriology
Description: Expectorated sputum or throat swab
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  A. xylososidans | 1 | 0
  MRSA | 0 | 0
  PA | 0 | 4
  Staph | 12 | 9
  Normal flora | 4 | 2
  PA and S. maltophilia | 0 | 0
  PA and Staph | 4 | 7
  Staph and A. xylososidans | 0 | 0
  S. maltophilia | 1 | 0

7. Secondary Outcome: Forced Vital Capacity
Description: Percent predicted of forced vital capacity.
Time Frame: 6 months
Population: PFT's not done on children under age of 5.
Measure: Mean (Standard Deviation); unit: Percent Predicted
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 11 | 9
Percent Predicted | 92.3 (7.3) | 83.9 (8.2)

8. Secondary Outcome: FEV1
Description: Forced expiratory volume at one second, percent predicted.
Time Frame: 6 months
Population: PFT's not done on children under age of 5.
Measure: Mean (Standard Deviation); unit: Percent predicted
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 11 | 9
Percent predicted | 81.5 (4.9) | 71.6 (8.3)

9. Secondary Outcome: C-Reactive Protein (CRP)
Description: CRP was measured to determine if this test fell during the course of treatment.
Time Frame: 6 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
milligrams per liter | 10.9 (5.6) | 14.7 (6.5)

10. Primary Outcome: BMI Percentile
Description: Body Mass Index percentile adjusted for sex and age. Not available for participants under 2 years of age.
Time Frame: 6 months
Population: All old enough to have BMI percentile calculated. BMI percentile not available for children under 2 years of age
Measure: Mean (Standard Deviation); unit: Percentile adjusted for age and sex
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 20 | 20
Percentile adjusted for age and sex | 47.5 (14.0) | 36.0 (17.0)

11. Secondary Outcome: White Blood Cell Count
Description: White blood cell count was measure at the beginning and end of the study to determine if treatment affected this test.
Time Frame: 6 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: 1000 cells/mm^3
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
1000 cells/mm^3 | 8.4 (1.5) | 9.5 (2.4)

12. Secondary Outcome: Vitamin E
Description: Serum Vitamin E levels were measured to determine if treatment affected this test.
Time Frame: 6 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: milligrams per liter
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
milligrams per liter | 8.6 (1.6) | 6.8 (1.4)

13. Primary Outcome: Weight Percentile
Description: Weight percentile, adjusted for sex and age
Time Frame: 6 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: Percentile adjusted for age and sex
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
Percentile adjusted for age and sex | 43.2 (12.3) | 31.8 (14.0)

14. Primary Outcome: Height Percentile
Description: The subjects were measured over the course of the study to determine if treatment improved height percentile.
Time Frame: 6 Months
Population: All participants.
Measure: Mean (Standard Deviation); unit: Percentile adjusted for age and sex
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
Percentile adjusted for age and sex | 43.3 (12.5) | 36.5 (13.2)

15. Primary Outcome: Fecal Calprotectin
Description: Fecal Calprotectin, a measure of gut inflammation, was measured to see if the treatment decreased this outcome.
Time Frame: 6 months
Population: All participants.
Measure: Mean (Standard Deviation); unit: Micrograms/gram feces
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
Micrograms/gram feces | 61.2 (26.4) | 76.6 (30.7)

16. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: ALT was measured to determine if liver function was affected by treatment over the course of the study.
Time Frame: 6 Months
Population: All participants.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Number analyzed (Participants) | 22 | 22
units per liter | 18.1 (7.0) | 25.8 (10.9)

17. Secondary Outcome: Bacteriology
Description: Expectorated sputum or throat swab
Time Frame: 6 Months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  A. xylososidans | 0 | 0
  MRSA | 0 | 1
  PA | 1 | 7
  Staph | 12 | 8
  Noraml flora | 6 | 0
  PA and S. maltophilia | 0 | 0
  PA and Staph | 1 | 5
  Staph and A. xylososidans | 0 | 0
  S. maltophilia | 1 | 1
  Strep B | 1 | 0

18. Secondary Outcome: Frequency of Abdominal Pain
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 15 | 9
  2- rare | 6 | 7
  3- frequently | 1 | 6
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

19. Secondary Outcome: Severity of Abdominal Pain
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 14 | 9
  2- light | 7 | 9
  3- moderate | 0 | 3
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

20. Secondary Outcome: Frequency of Belching
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 18 | 11
  2- rare | 4 | 6
  3- frequently | 0 | 5
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

21. Secondary Outcome: Severity of Belching
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 18 | 11
  2- light | 3 | 6
  3- moderate | 0 | 4
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

22. Secondary Outcome: Frequency of Flatulence
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 7 | 3
  2- rare | 14 | 10
  3- frequently | 1 | 9
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

23. Secondary Outcome: Severity of Flatulence
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 7 | 3
  2- light | 13 | 11
  3- moderate | 1 | 7
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

24. Secondary Outcome: Frequency of Lack of Appetite
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 11 | 4
  2- rare | 11 | 14
  3- frequently | 0 | 4
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

25. Secondary Outcome: Severity of Lack of Appetite
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 11 | 3
  2- light | 10 | 14
  3- moderate | 0 | 4
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

26. Secondary Outcome: Frequency of Bloating
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 6 | 2
  2- rare | 14 | 9
  3- frequently | 2 | 10
  4- constantly | 0 | 1
  Did Not Answer | 0 | 0

27. Secondary Outcome: Severity of Bloating
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 6 | 2
  2- light | 14 | 11
  3- moderate | 1 | 7
  4- serious | 0 | 1
  Did Not Answer | 1 | 1

28. Secondary Outcome: Frequency of Nausea
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 14 | 14
  2- rare | 8 | 7
  3- frequently | 0 | 1
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

29. Secondary Outcome: Severity of Nausea
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 13 | 13
  2- light | 8 | 7
  3- moderate | 0 | 1
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

30. Secondary Outcome: Frequency of Vomiting
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 21 | 15
  2- rare | 1 | 7
  3- frequently | 0 | 0
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

31. Secondary Outcome: Severity of Vomiting
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 20 | 14
  2- light | 1 | 7
  3- moderate | 0 | 0
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

32. Secondary Outcome: Frequency of Heart Burn
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 17 | 18
  2- rare | 5 | 3
  3- frequently | 0 | 1
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

33. Secondary Outcome: Severity of Heart Burn
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 17 | 18
  2- light | 4 | 2
  3- moderate | 0 | 1
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

34. Secondary Outcome: Frequency of Diarrhea
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 18 | 11
  2- rare | 4 | 8
  3- frequently | 0 | 3
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

35. Secondary Outcome: Severity of Diarrhea
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 17 | 10
  2- light | 4 | 8
  3- moderate | 0 | 3
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

36. Secondary Outcome: Frequency of More Than 2 Bowel Movements Per Day
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 15 | 12
  2- rare | 6 | 3
  3- frequently | 1 | 7
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

37. Secondary Outcome: Severity of More Than 2 Bowel Movements Per Day
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 14 | 12
  2- light | 7 | 4
  3- moderate | 0 | 5
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

38. Secondary Outcome: Frequency of Less Than 2 Bowel Movements Per Week
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most frequent
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- never | 19 | 16
  2- rare | 3 | 5
  3- frequently | 0 | 1
  4- constantly | 0 | 0
  Did Not Answer | 0 | 0

39. Secondary Outcome: Severity of Less Than 2 Bowel Movements Per Week
Description: Part of the Qualitative Symptom Assessment; scaled from 1-4 with 4 being the most severe
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Oral Reduced L-glutathione | Placebo Oral Calcium Citrate
Number analyzed (Participants) | 22 | 22
participants
  1- absent | 17 | 15
  2- light | 4 | 4
  3- moderate | 0 | 2
  4- serious | 0 | 0
  Did Not Answer | 1 | 1

ADVERSE EVENTS:
Time Frame: 6 months of the trial
Description: Patients kept a daily journal. They reported change in symptoms such as bloating, abdominal pain, as well as anorexia and hunger.
Arm/Group | Oral Reduced L-glutathione | Placebo Calcium Citrate
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
This trial was limited to one site. The number was relatively small. Since PFT's were not done on children under the age of 5, there is even smaller number of participants contributing PFT data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No